CLINICAL TRIAL: NCT05381324
Title: Fistula-associated Anal Adenocarcinoma - a Twenty Years' Single-center Experience.
Brief Title: Fistula-associated Anal Adenocarcinoma
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Felix Harpain, Dr.med.univ., Medical University of Vienna
Other Study IDs: 1258
Record Dates: First submitted 2022-05-14; First posted 2022-05-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The fistula-associated anal adenocarcinoma is rare in patients suffering from anal fistulas. There is only little data available for this patient collective making characterization and management of this disease difficult. Late diagnosis and advanced tumor stage at diagnosis result in poor clinical outcome. It is the purpose of this study to evaluate patients clinically diagnosed with a FAAC and to further perform a histopathological characterization of the available tumor specimen.

DETAILED DESCRIPTION:
All patients receiving surgery for an anal fistula in the years 1999 to 2019 at a tertiary university referral hospital were included in the analysis. A retrospective review of patients' charts was performed. Patients suffering from FAAC were eligible for histopathological analysis including immunohistochemistry and molecular profiling.

ELIGIBILITY:
Inclusion Criteria:

* anal fistula

Exclusion Criteria:

* previous cancer of the anal canal

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all patients receiving surgery for an anal fistula at a tertiary university referral hospital. Of those, patients suffering from fistula-associated anal cancer were eligible for further clinical and histopathological analysis
Sampling Method: Probability Sample
Enrollment: 1004 (Actual)
Dates: Start 1999-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
fistula-associated anal adenocarcinoma (FAAC) | 1999-2019
  include and analyze all patients suffering from FAAC

IPD SHARING:
Plan to Share IPD: No